CLINICAL TRIAL: NCT02705586
Title: Video Based Mindfulness Based Stress Reduction
Acronym: vMBSR
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Oregon Health and Science University (Other)
Collaborators: Portland VA Medical Center (U.S. Federal Agency)
Responsible Party: Principal Investigator, Amie Hiller, MD, Principal Investigator, Oregon Health and Science University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 15421; 3825 (Other: VA Portland Health Care System); 5410 (Other: Oregon Clinical and Translational Institute)
Record Dates: First submitted 2016-03-07; First posted 2016-03-10 (Estimated); Results first posted 2019-10-31 (Actual); Last update posted 2019-10-31 (Actual); Status verified 2019-10

CONDITIONS: Parkinson's Disease
Keywords: Movement disorders; Metabolic Stress
MeSH Terms: conditions — Parkinson Disease; Movement Disorders | interventions — Mindfulness; Mindfulness-Based Stress Reduction

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- only one arm - open label study (Experimental): 2 hour video based mindfulness-based stress reduction class once a week for 10 weeks.
  Interventions: Behavioral: Mindfulness

INTERVENTIONS:
Behavioral: Mindfulness — Mindfulness focuses on helping participants understand their personal reactions to stress, teaches skills that provide means to modify stress reactions, and promotes self-care and feelings of competence and mastery. In addition to weekly class sessions, participants are asked to do an hour of home practice the days that the class does not meet.
  Other Names: Mindfulness Based Stress REduction

SUMMARY:
To evaluate the feasibility of a video based mindfulness intervention for stress reduction and to evaluate the cortisol response in persons with PD and their caregivers. The data from this project will be used for a future grant application of a stress reduction intervention in persons with PD.

DETAILED DESCRIPTION:
Participants will be enrolled at the VA Portland and have a baseline assessment. The baseline will assess neurological disorders (including Parkinsonism) and current stress. All participants will attend 10 weeks of mindfulness based stress reduction (MBSR) through video feed on the Portland VA campus. During the week prior to the first class and the week after the last class, participants will complete questionnaires regarding stress, collect saliva samples, and, for the Parkinson's patient, monitor motor symptoms of PD using diaries and inertial sensors. A final visit will assess stress, neurological diseases, and Parkinsonism.

ELIGIBILITY:
Inclusion Criteria:

* Parkinson's disease
* Some Postural instability
* Tremor in upper limb
* Caregiver willing to also participate

Exclusion Criteria:

* No neurological disease
* Cognitive deficits
* Other neurological/psychological disorder
* Completion of a stress reduction program in the last 12 months

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2016-03; Primary Completion 2016-07 (Actual); Study Completion 2016-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Amie L Hiller (Peterson), MD, Principal Investigator — VA Porltand Health Care system
Locations (2):
- United States (2):
  - Oregon Health & Science University, Portland, Oregon
  - VA Portland Health Care System, Portland, Oregon

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Armento ME, Stanley MA, Marsh L, Kunik ME, York MK, Bush AL, Calleo JS. Cognitive behavioral therapy for depression and anxiety in Parkinson's disease: a clinical review. J Parkinsons Dis. 2012;2(2):135-51. doi: 10.3233/JPD-2012-12080. PMID 23939438
- [Result] Achey M, Aldred JL, Aljehani N, Bloem BR, Biglan KM, Chan P, Cubo E, Dorsey ER, Goetz CG, Guttman M, Hassan A, Khandhar SM, Mari Z, Spindler M, Tanner CM, van den Haak P, Walker R, Wilkinson JR; International Parkinson and Movement Disorder Society Telemedicine Task Force. The past, present, and future of telemedicine for Parkinson's disease. Mov Disord. 2014 Jun;29(7):871-83. doi: 10.1002/mds.25903. Epub 2014 May 17. PMID 24838316
- [Result] Almeida DM, Wethington E, Kessler RC. The daily inventory of stressful events: an interview-based approach for measuring daily stressors. Assessment. 2002 Mar;9(1):41-55. doi: 10.1177/1073191102091006. PMID 11911234

RESULTS

PARTICIPANT FLOW:
Recruitment Details: From March 2016 to May 2016, 8 Parkinson's disease veterans and their caregivers were recruited for the 10-week Mindfulness-Based Stress Reduction classes held at the VA Portland Health Care System in Portland, Oregon.
Pre-assignment Details: 13 participants consented for the study. 4 withdrew after screening prior to the intervention due to the amount of travel to the Portland VA in the study.
Period: Overall Study
Arm/Group | Only One Arm - Open Label Study
Started | 13
Completed | 5
Not Completed | 8
Not completed — Health Issues | 2
Not completed — Transportation Difficulties | 5
Not completed — Vacation/Planned Absence | 1

BASELINE CHARACTERISTICS:
Population: Baseline visits completed on 13 participants; Parkinson's disease and caregivers. 4 individuals dropped out prior to class week 1 due to difficulty travelling to the VA/too busy to come to the VA weekly. Analysis on 13 (individuals - both Parkinson's disease and caregivers).
Arm/Group | Only One Arm - Open Label Study
Number analyzed (Participants) | 13
Age, Continuous [Mean (Standard Deviation); unit: years] | 71.7 (6.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6
  Male | 7
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 13
Years of Formal Education [Mean (Standard Deviation); unit: years] | 14.9 (2.5)
Montreal Cognitive Assessment (MoCA) [Mean (Standard Deviation); unit: units on a scale] — The MoCA is a short cognitive screening test designed to assist health care professionals for the detection of mild cognitive impairment. The MoCA assesses cognitive function across a variety of domains, such as visuospatial /executive functioning, naming (animals), memory, attention, language, abstraction, delayed recall, and orientation. The MoCA is scored on a 0 to 30 scale, with lower numbers indicating more cognitive impairment. Scores ranging from 26 - 30 are normal, 18 - 26 mild impairment, 10 - 17 moderate impairment, and less than 10 severe cognitive impairment.
  units on a scale | 25.4 (2.2)
United Parkinsons Disease Rating Scale - Part III motor section (UPDRS) [Mean (Standard Deviation); unit: units on a scale] — This is the motor subsection of the UPDRS and is a commonly used tool to rate the symptoms of Parkinson's disease. Each item on the scale is rated from 0 (normal) to 4 (Can barely perform the task) several motor areas including speech, facial expression, tremor, rigidity, hand movements, agility, posture, and gait. Total score ranges from 0 to 108 with higher values on this scale represent a more severe stage of the disease. Population: 8/13 participants had Parkinson's disease. This questionnaire is only appropriate for Parkinson's disease participants.
  units on a scale
    number analyzed (Participants) | 8
    (all) | 26.6 (8.5)
Hoehn & Yahr [Mean (Standard Deviation); unit: units on a scale] — This is an objective staging scale for rating the clinical functioning of Parkinson's disease patients, combining functional deficits (disability) and objective signs (impairment). This staging scale is commonly used in both research settings and clinical practice. The Hoehn & Yahr is an ordinal scale ranging from 0 (no signs of disease) to 5 (wheelchair bound/bedridden). The modified version of the scale includes increments of 0.5. The HY has shown good inter-rater reliability and, although it is used worldwide, the clinimetric validity has not been established Population: 8/13 participants had Parkinson's disease. This questionnaire is only appropriate for Parkinson's disease participants.
  units on a scale
    number analyzed (Participants) | 8
    (all) | 2.2 (0.3)
Perceived Stress Scale (PSS) [Mean (Standard Deviation); unit: units on a scale] — The PSS consists of 10 questions rated on a scale of 0-4. A score of 40 would be the highest level of stress. A total score 13 was used as a cut-off point for stressed (>= 13) and less than 13 was categorized as non-stressed.
  units on a scale | 12.7 (7.5)
Hamilton Anxiety Rating Scale (HAM - A) [Mean (Standard Deviation); unit: units on a scale] — The HAM-A is a widely used measure of the severity of anxiety symptoms in adults, adolescents and children. The 14-item scale asks about a series of symptoms and measures both psychic anxiety (mental/psychological) and somatic anxiety (physical). Each item is scored on a scale of 0 (not present) to 4 (severe) with a total range 0-56. Greater than 17 indicates mild severity, 18-24 mild to moderate severity, and 25-30 moderate to severe.
  units on a scale | 10.8 (7.6)
Hamilton Depression Rating Scale (HAM - D) [Mean (Standard Deviation); unit: units on a scale] — The HAM-D is a widely used measure of the severity of depression. The HAM-D must be administered by a trained professional using a semi-structured interview. The HAM-D has been validated in a community sample of Parkinson's disease patients and has shown good convergent validity in de novo Parkinson's patients. Scoring is based on the first 17. Nine items are scored 0-2 with 0 indicating no difficulty. Eight items are scored on a 5-point scale ranging from 0 (not present) to 4 (severe). Scores range from 0 to 53 with higher scores indicating more severe depression.
  units on a scale | 7.2 (6.7)
Parkinson's Disease Questionnaire 39 (PDQ-39) [Mean (Full Range); unit: units on a scale] — The PDQ39 is a 39 item patient completed survey targeting well-being and functioning in PD. This scale address 8 dimensions (mobility, activities of daily living, emotional well-being, stigma, social support, cognitions, communication, and bodily discomfort). The dimension scores are on a scale of 0 ("Never") to 4 ("Always/Cannot Do"). Scale scores are summed and range from 0 to 100 with 100 being the maximum level of problems. The PDQ39 has shown adequate reliability and convergent validity. Population: 8 of the 13 participants had Parkinson's disease. This questionnaire is only appropriate for Parkinson's disease participants.
  units on a scale
    number analyzed (Participants) | 8
    (all) | 37.4 [16 to 75]
Parkinson Disease Questionnaire - Carer (PDQ-Carer) [Median (Full Range); unit: units on a scale] — This is a self-administered quality of life questionnaire specifically designed for the caregiver of a Parkinson's disease patient. The 29-item represents four discrete scales social and personal activities, anxiety and depression, self-care, and stress. All items are asked about the influence of caring on specific areas of life over the past four weeks and are rated on a 0 "Never" to 4 "Always" scale. Raw scores are summed and range from 0 to 100 with 100 being worst/maximum level of a problem. Population: 5/13 participants were caregivers of Parkinson's disease patients. This questionnaire is only appropriate for caregivers of Parkinson's disease participants. One participant did not complete the questionnaire because they were not in a caregiver role for the Parkinson's disease participant.
  units on a scale
    number analyzed (Participants) | 4
    (all) | 13 [6 to 27]

OUTCOME MEASURES:

1. Primary Outcome: Salivary Cortisol Levels (Pre- and Post-) Mindfulness-Based Stress Reduction Program
Description: Enzyme-linked immunoassay salivary cortisol levels (ng/mL) taken prior to Mindfulness-Based Stress Reduction will be compared to samples taken after the intervention.
Time Frame: Baseline to 12 weeks
Measure: Mean (Standard Deviation); unit: Concentration (ng/mL)
Arm/Group | Only One Arm - Open Label Study
Number analyzed (Participants) | 5
Concentration (ng/mL) | -33.1 (41.5)

ADVERSE EVENTS:
Arm/Group | Only One Arm - Open Label Study
Serious Adverse Events (participants affected / at risk) | 0/9
Other Adverse Events (participants affected / at risk) | 0/9

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes